CLINICAL TRIAL: NCT05969613
Title: Comparison of Regional Block, Wound Infiltration and Caudal Block for Post Operative Pain Management in Children Undergoing Inguinal Herniotomy
Brief Title: Comparison of Regional Block, Wound Infiltration and Caudal Block for Pain Management in Children
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fatima Numeri, Dr Fatima Naumeri Associate Professor, King Edward Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Fnaumeri
Record Dates: First submitted 2021-09-22; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regional Block (Experimental): Bupivacaine 0.25%
  Interventions: Procedure: Regional block
- Wound infilteration (Active Comparator): Bupivacaine 0.25%
  Interventions: Procedure: Wound infiltration
- caudal block (Active Comparator): Bupivacaine 0.25%
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Regional block — regional block with 0.25% Bupivacaine at a dose of 2ml/kg with adrenaline
  Arms: Regional Block
Procedure: Wound infiltration — Infiltration of surgical site with 0.25% Bupivacaine at 0.5ml/kg dose
  Arms: Wound infilteration
Procedure: Caudal block — Infiltration of caudal epidural space with 0.25% Bupivacaine at 1ml/kg dose
  Arms: caudal block

SUMMARY:
Comparison of regional block, wound infiltration and caudal block for post operative pain management in participants undergoing inguinal herniotomy.

DETAILED DESCRIPTION:
Investigators are comparing three modalities (regional block, wound infiltration and caudal block), for post operative pain management in participants after inguinal herniotomy.

ELIGIBILITY:
Inclusion Criteria:

1. •Patients under 13 years of age
2. •Inguinal hernia

Exclusion Criteria:

1. •History of allergy to any drugs used in study documented on history.
2. •Infection at the site of regional, caudal or local infiltration, documented on clinical examination.
3. •Irreducible, obstructed or strangulated hernia, documented on clinical examination.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
post operative pain -FLACC Pain sacle | Within 24 hours
  Post operative pain management will be calculated by use of FLACC Pain scale . An overall pain score ranging from 0 to 10.
post operative pain -Wong-Baker Faces pain scale | Within 24 hours
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Mamoonullah Asmati, Principal Investigator — King Edward Medical University
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan